CLINICAL TRIAL: NCT04284449
Title: Integrative Therapy for Holistic, Natural Cognition and Lifestyle Rehabilitation
Acronym: ITHNCLR
Status: Completed | Type: Observational
Sponsor: National University of Natural Medicine (Other)
Collaborators: North County Natural Medicine (Unknown)
Responsible Party: Principal Investigator, Ryan Bradley, Primary Investigator, National University of Natural Medicine
Other Study IDs: RB7102019
Record Dates: First submitted 2020-02-12; First posted 2020-02-25 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Cognitive Dysfunction
Keywords: Mild Cognitive Impairment (MCI); Cognitive Decline; Alzheimer's Disease (AD); Dementia
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease; Dementia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Enrolled Participants: This is a whole-practice precision medicine model in which a participant-specific Naturopathic treatment program is developed and implemented for older adults with cognitive complaints.
  Interventions: Other: Whole-practice cognitive optimization

INTERVENTIONS:
Other: Whole-practice cognitive optimization — This intervention is a whole-practice intervention that may include nutritional assessment & supplementation, determination of food sensitivities and dietary changes, natural products such as herbal anti-inflammatories, assessment of whole body-burden of toxicants (such as heavy metals and fungal toxins) and steps to reduce exposures, and behavioral changes such as exercise, meditation, and sleep hygiene optimization.

SUMMARY:
An observational study to determine outcomes of older adults who are under naturopathic medical care for cognitive complaints at a specific clinic in Southern California.

DETAILED DESCRIPTION:
This prospective observational study will examine patient outcomes associated with individualized, whole-system integrative medical care, provided by a naturopathic physician at a specific clinic in the state of California. Participants will be older adult patients of the clinic who present with objectively measurable cognitive dysfunction, and who elect to voluntarily participate in the study.

Participants' cognitive function will be assessed using validated objective (NIH Toolbox) and subjective (NIH Neuro-Quality of Life questionnaires) instruments. The primary outcomes are change from baseline to six months post-baseline in these two instruments.

Additionally, physical activity and sleep data will be tracked using wearable telemetry, and neurophysiological parameters will be measured with electroencephalography. Detailed treatment descriptions and adverse events will be tracked.

ELIGIBILITY:
Inclusion Criteria:

* Community-dwelling adults ≥60 years of age.
* Montreal Cognitive Assessment (MoCA) score of 12-23.
* Able to independently make decisions.
* Able to safely travel to North County Natural Medicine for 4 study visits and approximately 4 clinical visits, for a duration of 6 months.
* Able to wear an Oura Ring, download data every 6 days, and keep the ring regularly charged for the duration of participants' involvement in the study.
* A high school diploma or equivalent.
* Ability to communicate via email.
* Ability to independently fill out a computer-administered questionnaire.
* Ability to withhold from seeing another integrative or alternative medicine provider for the 6 months of participation in the study.

Exclusion Criteria:

* Inability to read and write in English.
* MoCA score >23.
* A visual impairment that would prevent reading a computer screen.
* Partial or full deafness.
* A previous diagnosis of dementia (e.g. Alzheimer's Disease or any other kind of dementia).
* Congenital cognitive impairment or disability.
* Alcohol or substance abuse.
* Serious somatic disease, neurodegenerative disease, acute onset of cognitive decline, or rapid neurological impairment.
* Inability to bring an affiliate to the Informed Consent Consultation.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy adults aged 60 years or more, with objectively measurable cognitive impairment, who volunteer to receive care at a specific clinic in Southern California.
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2020-02-24 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
NIH Toolbox-Cognitive Battery | Baseline, 6 months
  Change from baseline to 6 months in scores on a computer-administered cognitive function test
Quality of Life in Neurological Disorders questionnaire (Neuro-QoL) | Baseline, 6 months
  Change from baseline to 6 months in scores on a brief, validated questionnaire that monitors the physical, mental, and social effects experienced by individuals living with neurological conditions

SECONDARY OUTCOMES:
Event-related potential (P300) | 6 months post-baseline visit
  Change from baseline to 6 months of an auditory event provoked change in electrical potential of the brain, measured noninvasively by electroencephalography (EEG)
Peak alpha frequency | 6 months post-baseline visit
  Change from baseline to 6 months of the peak (highest intensity) frequency in electrical activity of the brain between 8 Hz and 12 Hz, measured noninvasively by electroencephalography (EEG)
Physical activity | 6 months
  Change from baseline to 6 months in participants' overall physical activity as measured with telemetry from a wrist-worn activity tracker
Sleep quantity | 6 months
  Change from baseline to 6 months in participants' total sleep as measured with telemetry from a wrist-worn activity tracker
Number and type of Adverse Events | From enrollment through study completion, a period of 6 months
  Total number of adverse events and serious adverse events (using NIH's Common Terminology Criteria for Adverse Events version 4.0)

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Bradley, ND, Principal Investigator — National University of Natural Medicine; Heather Sandison, ND, Principal Investigator — North County Natural Medicine
Locations (1):
- North County Natural Medicine, Encinitas, California, United States

IPD SHARING:
Plan to Share IPD: No